CLINICAL TRIAL: NCT02794129
Title: Functional Magnetic Resonance Imaging of Formal Thought Disorders in Bipolar Disorder
Brief Title: fMRI of Flight of Ideas in Bipolar Disorder
Acronym: i-TCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PJ12075
Record Dates: First submitted 2016-05-30; First posted 2016-06-08 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2016-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

ARMS (2):
- Bipolar Disorder patients (Experimental)
  Interventions: Other: Functional Magnetic Resonance Imaging
- Healthy Controls (Experimental)
  Interventions: Other: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging

SUMMARY:
Bipolar disorder is a mental disease characterized by mood dysregulation and arises from manic, depressive or mixed episodes. The observations of the patient's speech and language behaviour due to flight of ideas or loss of goal probably result from an underlying disturbance in semantic networks dealing with semantic associations. The aim of our study will be to have a better comprehension of thought disorders in bipolar disorder by cognitive exploration of semantic processing.

DETAILED DESCRIPTION:
Bipolar disorder is a mental disease characterized by mood dysregulation and arises from manic, depressive or mixed episodes. During these episodes, formal thought disorders are observed, associated to emotional perturbation, behaviour troubles and some psychotic symptoms. During mania, the type of thought disorders observed are derailment, flight of ideas, with an increase in the amount of spontaneous speech and loss of goal. These observations of the patient's speech and language behaviour probably result from an underlying disturbance in semantic networks dealing with semantic associations. These networks have been studied extensively in schizophrenia but remain unknown in bipolar disorder. In this context, the aim of our study will be to have a better comprehension of formal thought disorders in bipolar disorder by cognitive exploration of semantic activation and inhibition.

ELIGIBILITY:
Inclusion criteria

BD patients :

* Men or women, right-handed
* diagnosis of type 1 bipolar disorder, according to the DSM-IV criteria
* aged from 18 to 65 years-old
* Native French speaker
* Affiliated to the social security

Healthy Controls (HC):

* Men or women, right-handed
* aged from 18 to 65 years-old
* Native French speaker
* Affiliated to the social security

Exclusion criteria

BD patients :

* recent alcohol and/or drug abuse or dependence
* significant general medical illness, including neurological disorders or head trauma
* sensorial impairment (visual and/or hearing)
* Contraindication to the use of MRI

HC:

* first-degree-relative history of bipolar disorder, schizophrenia or schizoaffective disorder according to DSM-IV
* recent alcohol and/or drug abuse or dependence
* significant general medical illness, including neurological disorders or head trauma
* sensorial impairment (visual and/or hearing)
* Contraindication to the use of MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
brain activation profiles by Functional Magnetic Resonance Imaging | inclusion visit

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] Raucher-Chene D, Terrien S, Gierski F, Obert A, Caillies S, Besche-Richard C, Kaladjian A. Neural Correlates of Semantic Inhibition in Relation to Hypomanic Traits: An fMRI Study. Front Psychiatry. 2018 Apr 4;9:108. doi: 10.3389/fpsyt.2018.00108. eCollection 2018. PMID 29670548